CLINICAL TRIAL: NCT07143279
Title: Testosterone Supplementation in Patients in Best Supportive Care: Impact on Quality of Life
Acronym: TestoSup
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-SP01-2025; 2025-522023-10-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-03; First posted 2025-08-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hypotestosteronism; Palliative Care
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testosterone supplementation in patients in best supportive care: impact on quality of life (Experimental): Single-arm prospective pilot study that will enrol hypogonadal (testosterone < 231 ng/dL) male subjects in best supportive care, with no further therapeutic options and no need for resuscitation.
  Administration of Sustanon 250® (1 ml, IM) on day 0 after confirmation of hypogonadism by blood test and then every 15 days.
  Interventions: Drug: Sustanon 250

INTERVENTIONS:
Drug: Sustanon 250 — Sustanon 250® (1 ml, IM) every 10 days
  Other Names: Testosterone

SUMMARY:
This is a monocentric, single-arm prospective pilot study that will enrol hypogonadal (testosterone < 231 ng/dL) male subjects in best supportive care, with no further therapeutic options and no need for resuscitation.

Currently, testosterone formulations for intramuscular (IM) injection and subcutaneous injection as well as for oral and transdermal administration have been approved for androgen therapy. To date, injectable testosterone is the most commonly used formulation. To increase serum testosterone levels to the physiological range IM injections of testosterone every 2-3 weeks are required, which lead to supraphysiological peaks shortly after administration, followed by a sharp fall in levels thereafter. Testosterone levels before the next injection are frequently in the hypogonadal range. For this reason, Sustanon 250® (1 ml, IM) will be administered on day 0 after confirmation of hypogonadism by blood test and then every 15 days in this trial given the limited life expectancy of the subjects and to maximise the effect and benefit of testosterone supplementation.

The Edmonton questionnaire and ADL questionnaire will be completed before the injection on day 0 and then every 15 days at the time of injection until subject's death or if a subject is discontinued from the study treatment/procedures for any other reasons than death. In parallel, the EQ-5D-3L questionnaire will be completed by a family member or a proxy.

ELIGIBILITY:
Inclusion Criteria:

1. Male hypogonadal with total testosterone < 231 ng/dl in best supportive care with no further therapeutic options and who do not wish to be reanimated.
2. Age ≥ 18 years old
3. Patient able to understand the patient information sheet and able to sign the Informed Consent form (ICF) prior to any study related procedure.

Exclusion Criteria:

1. Untreated prostate cancer, given the risk of epiduritis.
2. Known hypersensitivity reactions to the study drug or to any excipients.
3. Known allergies to peanuts or soya.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessed by ADL questionnaire | Every 15 days through study completion
  Best improvement over time in independence using the ADL independence scale in terms of personal hygiene, dressing, going to the toilet, locomotion, continence and eating.
  The primary endpoint is defined as the difference between the best score after baseline and the initial score at baseline.
Quality of life assessed by Edmonton Symptom Assessment Scale | Every 15 days through study completion,
  Best improvement over time in symptoms of pain, fatigue, sadness, anxiety, drowsiness, appetite, sense of well-being, shortness of breath, bowel movements and strength using the Edmonton Symptom Assessment Scale.
  The primary endpoint is defined as the difference between the best score after baseline and the initial score at baseline.

SECONDARY OUTCOMES:
EQ-5D-3L questionnaire | Every 15 days through study completion
  Improvement of quality of life of subjects from the point of view of a proxy using the EQ-5D-3L questionnaire (EQ-5D-3L scale 0-100 where 0=worst outcome and 100=better outcome)
Dynamic/change of the ADL and Edmonton System Assessment Scale during treatment | At each time point during treatment, especially at Day 15.
  The average of ADL and Edmonton Symptom Assessment Scale during treatment after baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium